CLINICAL TRIAL: NCT00702234
Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established After Controlled Ovarian Stimulation in Clinical Trial 38825 for Org 36286 (Corifollitropin Alfa)
Brief Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established in Clinical Trial P05714 (Care Program)(P05715)
Acronym: Care
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05715; 2004-004967-30 (EudraCT Number); 38829 (Other: Organon); MK-8962-008 (Other: Merck)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy; Neonates
Keywords: Neonatal outcome; Congenital malformations; In-Vitro fertilization; Controlled ovarian stimulation; Follow-up
MeSH Terms: conditions — Congenital Abnormalities | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Progesterone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women/Expectant Mothers - Corifollitropin Alfa 150 µg: In base study P05714 (NCT00696878), up to 3 COS cycles were performed, each including the following: A single injection of 150 µg corifollitropin alfa was administered on Day 2 or 3 of the menstrual cycle (Stimulation Day 1). Administration of Gonadotropin Releasing Hormone (GnRH) antagonist (0.25 mg/day) started on Stimulation Day 5 or 6 and continued through day of administration of recombinant Human Chorion Gonadotropin ([rec]hCG) (5,000-10,000 IU/250 µg). Daily dosing with Follicle Stimulating Hormone (FSH) (not to exceed 225 IU/day) began on Stimulation Day 8 and continued up to day of (rec)hCG administration. Progesterone was administered for luteal phase support. After COS cycles 1 and 2, Frozen-Thawed Embryo Transfer cycles (up to 3 after each COS cycle) could occur. Participants with confirmed pregnancy at least 10 weeks after fresh embryo transfer in the base study were eligible for this follow-up study. In this follow-up study P05715, no study drugs were administered.
  Interventions: Biological: Corifollitropin alfa; Biological: GnRH antagonist; Biological: (rec)hCG; Biological: FSH; Drug: Progesterone

INTERVENTIONS:
Biological: Corifollitropin alfa — Subcutaneous (SC) administration of corifollitropin alfa at a dose of 150 μg in base study P05714 (NCT00696878). In this follow-up study P05715, no study medications were administered.
  Other Names: Org 36286; SCH 900962; MK-8962
Biological: GnRH antagonist — SC administration of a GnRH antagonist at a dose of 0.25 mg/day in base study P05714 (NCT00696878). In this follow-up study P05715, no study medications were administered.
Biological: (rec)hCG — SC administration of (rec)hCG at a dose of 5,000-10,000 IU/250 µg in base study P05714 (NCT00696878). In this follow-up study P05715, no study medications were administered.
Biological: FSH — SC administration of FSH at a dose not to exceed 225 IU/day in base study P05714 (NCT00696878). In this follow-up study P05715, no study medications were administered.
Drug: Progesterone — Vaginal administration of progesterone at a dose of at least 600 mg/day in base study P05714 (NCT00696878). In this follow-up study P05715, no study medications were administered.

SUMMARY:
The objective of this trial is to evaluate whether corifollitropin alfa (Org 36286) treatment for the induction of multifollicular growth in women undergoing controlled ovarian stimulation (COS) prior to in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) is safe for pregnant participants and their offspring. In addition, a primary efficacy variable, live birth rate, was evaluated.

DETAILED DESCRIPTION:
This is a follow-up protocol to prospectively monitor pregnancy, delivery, and neonatal outcomes of women who were treated with corifollitropin alfa and became pregnant after fresh embryo transfer during the base study P05714 (NCT00696878). For this trial, no study specific assessments are required, but information as obtained in standard practice will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in base study P05714 (NCT00696878) and received at least one dose of corifollitropin alfa in base study P05714;
* Ongoing pregnancy confirmed by ultrasound at least 10 weeks after a fresh embryo transfer in base study P05714;
* Able and willing to give written informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with an ongoing pregnancy at least 10 weeks after fresh embryo transfer in base study P05714 (NCT00696878) were enrolled in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2007-02-15 (Actual); Primary Completion 2009-10-22 (Actual); Study Completion 2010-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Bonduelle M, Mannaerts B, Leader A, Bergh C, Passier D, Devroey P. Prospective follow-up of 838 fetuses conceived after ovarian stimulation with corifollitropin alfa: comparative and overall neonatal outcome. Hum Reprod. 2012 Jul;27(7):2177-85. doi: 10.1093/humrep/des156. Epub 2012 May 15. PMID 22587997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 272 participants with ongoing pregnancy at 10 weeks after fresh embryo transfer (ET) in base study P05714 (NCT00696878), 268 enrolled in this follow-up study P05715. A participant could enter follow-up study without meeting formal definition for "Completion" of base study.
Pre-assignment Details: To complete base study P05714 (NCT00696878), a participant must have embryo transfer in the 3rd Controlled Ovarian Stimulation (COS) cycle (Treatment Cycle 3). For this follow-up trial P05715, study completion for participant (expectant mother) or live born infant was defined as completion of infant follow-up visit at 4-12 weeks after delivery.
Groups:
- Women/Expectant Mothers - Corifollitropin Alfa 150 µg: In base study P05714 (NCT00696878), up to 3 COS cycles were performed, each including the following treatments: A single injection of 150 µg corifollitropin alfa was administered on Day 2 or 3 of the menstrual cycle (Stimulation Day 1). Administration of Gonadotropin Releasing Hormone (GnRH) antagonist (0.25 mg/day) started on Stimulation Day 5 or 6 and continued through day of administration of recombinant Human Chorion Gonadotropin ([rec]hCG) (5,000-10,000 IU/250 µg). Daily dosing with Follicle Stimulating Hormone (FSH) (not to exceed 225 IU/day) began on Stimulation Day 8 and continued up to day of (rec)hCG administration. Progesterone was administered for luteal phase support. After COS cycles 1 and 2, Frozen-Thawed Embryo Transfer cycles (up to 3 after each COS cycle) could occur. Participants with confirmed pregnancy at least 10 weeks after fresh ET in the base study were eligible for this follow-up study. In this follow-up study P05715, no study drugs were administered.
- Fetuses Present at 10 Weeks After Fresh ET in Base Study: This group includes fetuses associated with expectant mothers who were administered corifollitropin alfa in base study P05714 (NCT00696878) who were enrolled in this follow-up study P05715. The fetuses were present at 10 weeks after fresh ET in base study P05714 and/or at enrollment of the expectant mother in this follow-up study P05715.
Period: Base Study (NCT00696878)
Arm/Group | Women/Expectant Mothers - Corifollitropin Alfa 150 µg | Fetuses Present at 10 Weeks After Fresh ET in Base Study
Started | 682 | 0
Completed | 178 | 0
Not Completed | 504 | 0
Period: Follow-up Study: Expectant Mothers
Arm/Group | Women/Expectant Mothers - Corifollitropin Alfa 150 µg | Fetuses Present at 10 Weeks After Fresh ET in Base Study
Started | 268 (A participant could enter follow-up study without meeting definition for "Completion" of base study) | 0
Completed | 246 | 0
Not Completed | 22 | 0
Period: Follow-up Study: Fetuses/Infants
Arm/Group | Women/Expectant Mothers - Corifollitropin Alfa 150 µg | Fetuses Present at 10 Weeks After Fresh ET in Base Study
Started | 0 | 315 (Fetuses present 10 weeks after fresh ET and/or at enrollment of expectant mother in follow-up study)
Live Born Infants | 0 | 304 (Of the 11 that were not live born infants, outcome is known for 8 (fetus was lost) and unknown for 3)
Completed | 0 | 288 (All 288 who completed were live born infants)
Not Completed | 0 | 27

BASELINE CHARACTERISTICS:
Population: Individuals who participated in base study P05714 (NCT00696878) and received at least one dose of corifollitropin alfa, who had an ongoing pregnancy confirmed by ultrasound at least 10 weeks after fresh ET in base study P05714 and were able and willing to give written informed consent to be enrolled in the follow-up study.
Groups:
- Expectant Mothers - Corifollitropin Alfa 150 µg: In base study P05714 (NCT00696878), up to 3 COS cycles were performed, each including the following treatments: A single injection of 150 µg corifollitropin alfa was administered on Day 2 or 3 of the menstrual cycle (Stimulation Day 1). Administration of GnRH antagonist (0.25 mg/day) started on Stimulation Day 5 or 6 and continued through day of administration of (rec)hCG (5,000-10,000 IU/250 µg). Daily dosing with FSH (not to exceed 225 IU/day) began on Stimulation Day 8 and continued up to day of (rec)hCG administration. Progesterone was administered for luteal phase support. After COS cycles 1 and 2, Frozen-Thawed Embryo Transfer cycles (up to 3 after each COS cycle) could occur. Participants with confirmed pregnancy at least 10 weeks after fresh ET in the base study were eligible for this follow-up study. In this follow-up study P05715, no study drugs were administered.
Arm/Group | Expectant Mothers - Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With Ongoing Pregnancy After a Corifollitropin Alfa COS Cycle in Base Study and ≥1 Live Born Infant During Follow-up (Live Birth Rate)
Description: The live birth rate was defined as the number of participants who had an ongoing pregnancy after a corifollitropin alfa COS cycle in base study P05714 (NCT00696878) and who had at least one live born infant during follow-up, divided by the number of participants treated in the base study. For this analysis, it was assumed that any participants with ongoing pregnancy after a COS cycle in base study who did not enroll in follow-up study P05715 had no live born infants.
Time Frame: Up to approximately 32 months after first dose of corifollitropin alfa in base study P05714 (NCT00696878)
Population: Participants administered corifollitropin alfa in base study P05714 (NCT00696878)
Measure: Number; unit: percentage of participants
Groups:
- Women - Corifollitropin Alfa 150 µg: In base study P05714 (NCT00696878), up to 3 COS cycles were performed, each including the following treatments: A single injection of 150 µg corifollitropin alfa was administered on Day 2 or 3 of the menstrual cycle (Stimulation Day 1). Administration of GnRH antagonist (0.25 mg/day) started on Stimulation Day 5 or 6 and continued through day of administration of (rec)hCG (5,000-10,000 IU/250 µg). Daily dosing with FSH (not to exceed 225 IU/day) began on Stimulation Day 8 and continued up to day of (rec)hCG administration. Progesterone was administered for luteal phase support. After COS cycles 1 and 2, Frozen-Thawed Embryo Transfer cycles (up to 3 after each COS cycle) could occur. Participants with confirmed pregnancy at least 10 weeks after fresh ET in the base study were eligible for this follow-up study. In this follow-up study P05715, no study drugs were administered.
Arm/Group | Women - Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
percentage of participants | 37.8

2. Primary Outcome: Number of Expectant Mothers Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From approximately 10 weeks after fresh ET in base study P05714 up to birth of infant (up to approximately 6 months)
Population: Follow-up safety analysis was performed on expectant mothers who received corifollitropin alfa in base study P05714 (NCT00696878) and who enrolled in the follow-up study.
Measure: Number; unit: participants
Arm/Group | Expectant Mothers - Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 268
participants | 203

3. Primary Outcome: Number of Expectant Mothers Experiencing Serious AEs (SAEs)
Description: An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: From approximately 10 weeks after fresh ET in base study P05714 up to birth of infant (up to approximately 6 months)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Expectant Mothers - Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 268
participants | 145

4. Primary Outcome: Number of Live Born Infants Experiencing AEs
Description: as for outcome 2
Time Frame: Up to 12 weeks after birth
Population: Follow-up safety analysis was performed on live born infants delivered by expectant mothers who received corifollitropin alfa in base study P05714 (NCT00696878) and who enrolled in the follow-up study.
Measure: Number; unit: participants
Groups:
- Live Born Infants: This group includes infants born to mothers who were administered corifollitropin alfa in base study P05714 (NCT00696878) and who were enrolled in this follow-up study P05715. These infants, whose gestation outcome was live birth, are a subgroup of the total number of fetuses that were present at 10 weeks after fresh ET in base study P05714 and/or at enrollment of the expectant mother in this follow-up study P05715. Fetuses not born alive or with unknown outcome are not included in this reporting group.
Arm/Group | Live Born Infants
Number analyzed (Participants) | 304
participants | 99

5. Primary Outcome: Number of Live Born Infants Experiencing SAEs
Description: as for outcome 3
Time Frame: Up to 12 weeks after birth
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Live Born Infants
Number analyzed (Participants) | 304
participants | 79

ADVERSE EVENTS:
Time Frame: From approximately 10 weeks after fresh ET in base study P05714 (NCT00696878) up to 12 weeks after birth in current follow-up study (Up to approximately 9 months).
Arm/Group | Expectant Mothers - Corifollitropin Alfa 150 µg | Fetuses Present at 10 Weeks After Fresh ET in Base Study
Serious Adverse Events (participants affected / at risk) | 145/268 | 84/315
Other Adverse Events (participants affected / at risk) | 0/268 | 0/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expectant Mothers - Corifollitropin Alfa 150 µg (N=268) | Fetuses Present at 10 Weeks After Fresh ET in Base Study (N=315)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Disseminated intravascular coagulation in newborn (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia foetal (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia neonatal (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest neonatal (Cardiac disorders) | 0 (0) | 1 (1)
Foetal heart rate disorder (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Anal atresia (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Anomaly of external ear congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 4 (5)
Cleft palate (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital cytomegalovirus infection (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital hand malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital hydrocephalus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital infection (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital nose malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital pulmonary artery anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital pulmonary hypertension (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital tongue anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital torticollis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cystic lymphangioma (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Duodenal atresia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Dysmorphism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Factor IX deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Factor VIII deficiency (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Oculoauriculovertebral dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 5 (5)
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pulmonary malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pulmonary sequestration (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Renal dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Skull malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Solitary kidney (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Strabismus congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Syndactyly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Trisomy 18 (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 3 (3)
VACTERL syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 2 (2)
Retinopathy of prematurity (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 10 (10)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Neonatal infection (Infections and infestations) | 0 (0) | 2 (2)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 1 (1)
Uterine infection (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Perineal laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Amniotic fluid volume decreased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Foetal heart rate abnormal (Investigations) | 1 (1) | 0 (0)
Foetal heart rate increased (Investigations) | 1 (1) | 0 (0)
Gestational diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Delayed fontanelle closure (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage neonatal (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 4 (5) | 0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 18 (18) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Delayed delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Foetal acidosis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 0 (0)
Foetal growth retardation (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Foetal malposition (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 11 (11)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Multiple pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 0 (0)
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 50 (50)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 22 (22) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0)
Previous caesarean section (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 7 (7)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Twin pregnancy (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 0 (0)
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Perineal fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal laceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immature respiratory system (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (12)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 2 (2) | 0 (0)
Caesarean section (Surgical and medical procedures) | 3 (3) | 0 (0)
Selective abortion (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications must be based on data validated and released by the Sponsor. Any scientific paper, presentation, or other communication concerning the study must first be submitted to the Sponsor, at least 6 weeks prior to estimated publication or presentation, for written consent. Sponsor has the right to make its consent conditional upon proper representation of the interpretation of both the Sponsor and the Investigator in the discussion of the data in such communications.